CLINICAL TRIAL: NCT01990924
Title: Low Rate Fluoroscopy at Reducing Operator and Patient Radiation Dose During Transradial Coronary Diagnostic Angiography and Interventions
Brief Title: Low Rate Fluoroscopy to Reduce Radiation Dose During Coronary Angiography and Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, Study Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7.5 vs 15 Cine; 7.5 vs 15 (Other: ICICTA)
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Stable Angina; Unstable Angina; Acute Coronary Syndrome
Keywords: fluoroscopy; radiation; transradial; diagnostic; angiography; cardiac; coronary; angioplasty
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Acute Coronary Syndrome; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7.5 FPS (Experimental): Low rate fluoroscopy at 7.5 frames per second (FPS)
  Interventions: Radiation: 7.5 FPS
- 15 FPS (Active Comparator): Conventional rate fluoroscopy at 15 FPS
  Interventions: Radiation: 15 FPS

INTERVENTIONS:
Radiation: 15 FPS — X-ray pictures
  Other Names: Standard practice, conventional 15 frames per second (FPS)
  Arms: 15 FPS
Radiation: 7.5 FPS — X-ray pictures
  Other Names: Low rate fluoroscopy at 7.5 FPS
  Arms: 7.5 FPS

SUMMARY:
Objectives: To determine the efficacy of low rate fluoroscopy at 7.5 frames per second (FPS) vs. conventional 15 FPS for reduction of operator and patient radiation dose during diagnostic coronary angiography and percutaneous coronary intervention via the transradial approach.

Background: Transradial approach for cardiac catheterization is potentially associated with increased radiation exposure. Low rate fluoroscopy has potential to reduce radiation exposure.

DETAILED DESCRIPTION:
Methods: Patients undergoing transradial approach diagnostic angiography ± ad hoc PCI, wil be randomized to fluoroscopy at 7.5 FPS vs. 15 FPS prior to procedure. Both 7.5 and 15 FPS fluoroscopy protocols will be configured with a fixed dose per pulse of 40 nGy. Primary endpoints will be operator radiation dose (measured with dosimeter attached to the left side of thyroid shield in µSv), patient radiation dose (expressed as dose-area product in μGy.m2), and fluoroscopy time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective, urgent or emergent cardiac catheterization procedures with or without ad hoc PCI, via transradial approach are eligible.

Exclusion Criteria:

* 1) non-transradial access and 2) participation in research project(s) requiring higher ie 30 FPS cine angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Radiation Exposure | During Cardiac Catheterization
  Operator radiation dose (measured with dosimeter attached to the left side of thyroid shield, in µSv)
Radiation Exposure | During Cardiac Catheterization
  Patient radiation dose (expressed as dose-area product [DAP] in μGy.m2)
Radiation Exposure | During Cardiac Catheterization
  Fluoroscopy time

SECONDARY OUTCOMES:
Procedural Characteristics | During Cardiac Catheterization
  Procedural duration
Procedural Characteristics | During Cardiac Catheterization
  Total contrast volume used

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD PhD, Study Chair — International Chair on Interventional Cardiology and Transradial Approach
Locations (1):
- IUCPQ - Laval Hospital, Québec, Quebec, Canada

REFERENCES:
- [Derived] Abdelaal E, Plourde G, MacHaalany J, Arsenault J, Rimac G, Dery JP, Barbeau G, Larose E, De Larochelliere R, Nguyen CM, Allende R, Ribeiro H, Costerousse O, Mongrain R, Bertrand OF; Interventional Cardiologists at Quebec Heart-Lung Institute. Effectiveness of low rate fluoroscopy at reducing operator and patient radiation dose during transradial coronary angiography and interventions. JACC Cardiovasc Interv. 2014 May;7(5):567-74. doi: 10.1016/j.jcin.2014.02.005. Epub 2014 Apr 16. PMID 24746649